CLINICAL TRIAL: NCT01900262
Title: The Effects of Isolated Strengthening and Functional Training on Strength, Running Mechanics, Postural Control and Injury Prevention in Novice Runners
Brief Title: Exercise Interventions, Running Biomechanics and Injury in Novice Runners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: Biomechanigg Research Ltd. (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jennifer Baltich, Doctoral Student, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RRI2014
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Running; Leg Injuries
Keywords: Biomechanics; Ankle Strength; Postural Control; Running Mechanics
MeSH Terms: conditions — Leg Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strengthening (Experimental): Novice recreational runners from the Calgary area.
  Interventions: Other: Strengthening
- Balance Training (Experimental): Novice recreational runners from the Calgary area.
  Interventions: Other: Balance Training
- Stretching (Experimental): Novice recreational runners from the Calgary area.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Strengthening — Participants will be asked to complete 8 weeks of isolated ankle strengthening at home.
  Arms: Strengthening
Other: Balance Training — Participants will be asked to compete 8 weeks of functional balance training at home.
  Arms: Balance Training
Other: Stretching — Participants will be asked to complete a standard of practice static and dynamic stretching warm-up for 8 weeks at home.
  Arms: Stretching

SUMMARY:
The purpose of this study is to understand the effects of muscle strengthening and balance exercise interventions on muscle strength, running mechanics and postural control in novice recreational runners. Participants will be assessed before and after they engage in an 8-week exercise intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Novice recreational runners
* Less than one year of running experience
* Run at least twice a week for a total weekly distance between 5 and 15 km as your main form of physical activity
* 18-50 years of age

Exclusion Criteria:

* Neurological abnormalities or lower extremity injury or pain within three months of enrollment.
* No extensive history with balance training or isolated ankle strengthening within the last year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change in Strength | Week 0, Week 8
  Strength of the muscles crossing the ankle, knee and hip joint will be assessed at baseline and after 8 weeks of training in order to assess the change in strength following training.
Change in Running Mechanics | Week 0, Week 8
  Running kinematics and kinetics will be measured using 3D motion capture technology at baseline and after 8 weeks of training in order to assess the change in running mechanics following training.
Change in Postural Control | Week 0, Week 8
  Postural control will be assessed using single leg stance and the star excursion balance test at baseline and after 8 weeks of training in order to assess the change in postural control following training.

SECONDARY OUTCOMES:
Cumulative Running Related Injuries | Week 0 through Week 24
  Self-reported running-related injuries will be collected on a weekly basis for a total of 6 months following enrollment in order to quantify the cumulative amount of injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Baltich J, Emery CA, Whittaker JL, Nigg BM. Running injuries in novice runners enrolled in different training interventions: a pilot randomized controlled trial. Scand J Med Sci Sports. 2017 Nov;27(11):1372-1383. doi: 10.1111/sms.12743. Epub 2016 Aug 3. PMID 27486011
- [Derived] Baltich J, Emery CA, Stefanyshyn D, Nigg BM. The effects of isolated ankle strengthening and functional balance training on strength, running mechanics, postural control and injury prevention in novice runners: design of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Dec 4;15:407. doi: 10.1186/1471-2474-15-407. PMID 25471989